CLINICAL TRIAL: NCT00668460
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability, Dermical Sensitivity) of Dermacyd Delicata Pocket BR.
Brief Title: Dermatological Evaluation of Topic Compatibility-Dermacyd Delicata Pocket BR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: GMA-CO/Medical Director, sanofi-aventis administrative office France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_03744
Record Dates: First submitted 2008-04-23; First posted 2008-04-29 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lactic acid (Dermacid)

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermal irritability and cumulated dermal irritability) and allergy (sensibilization) of the product Dermacyd Pocket BR.

ELIGIBILITY:
Inclusion Criteria:

* Phototype Skin I,II, III e IV
* Integral skin test in the region

Exclusion Criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs
* Personnel history of atopy
* History of sensitivity or irritation for topic products
* Active cutaneous disease
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermal irritability and dermical sensitivity will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis administrative office, São Paulo, São Paulo, Brazil